CLINICAL TRIAL: NCT05493865
Title: Effects of Parent-Child Single-Session Growth Mindset Intervention on Adolescent Depression and Anxiety Problems: A Three-Arm Waitlist Randomised Controlled Trial
Brief Title: Parent-Child Single-Session Growth Mindset Intervention on Adolescent Depression and Anxiety Problems
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSEARS20211009001
Record Dates: First submitted 2022-08-07; First posted 2022-08-09 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-02

CONDITIONS: Depression, Anxiety
Keywords: implicit theory, fixed mindset, mental health, secondary school students, belief in change
MeSH Terms: conditions — Depression; Anxiety Disorders; Psychological Well-Being

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of intervention, blinding participants to the allocation is impossible. But Before the intervention starts, participants have no knowledge on which group they are belonging to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The Parent-Child Single-Session-intervention of Mindset Intelligence, Failure and Emotion (PC-SMILE) (Experimental): The PC-SMILE integrates the growth mindsets of intelligence, failure, and negative emotions and introduces these growth mindsets to students and parents, which consist of five components: (a) an introduction to brain functions regarding the potential of neuroplasticity and the possibility of changes in intelligence and emotions; (b) stories and testimonials from high-school-aged youths who describe their beliefs-in-change; (c) short videos with stories of improving intelligence and emotions and of failure-is-enhancing; (d) common questions and misconceptions about growth mindset; and (e) self-persuasion writing exercises in which the participants write notes to young students/others about the growth mindsets. The interventions for parents and students are different in terms of narrative and content. A total of 10 weekly booster messages with core intervention content will be sent between the two-week post-test and the three-month follow-up survey.
  Interventions: Behavioral: The Parent-Child Single-Session-intervention of Mindset Intelligence, Failure and Emotion (PC-SMILE)
- The Child Single-Session-intervention of Mindset Intelligence, Failure and Emotion (C-SMILE) (Experimental): The C-SMILE only provides intervention to children, which has the same components as PC-SMILE.
  Interventions: Behavioral: The Parent-Child Single-Session-intervention of Mindset Intelligence, Failure and Emotion (PC-SMILE)
- Waitlist control group (No Intervention): The waitlist control group will continue with normal education activities and do the pre- and post-intervention surveys at the same timeframe as the intervention groups. Participants in the waitlist group and C-SMILE group will be invited to complete the PC-SMILE after the three-month post-intervention survey.

INTERVENTIONS:
Behavioral: The Parent-Child Single-Session-intervention of Mindset Intelligence, Failure and Emotion (PC-SMILE) — This study will be a three-arm cluster-randomised controlled trial to examine the efficacy of the PC-SMILE for adolescents by comparing to a C-SMILE intervention group and a no-intervention waitlist control group.
  Arms: The Child Single-Session-intervention of Mindset Intelligence, Failure and Emotion (C-SMILE); The Parent-Child Single-Session-intervention of Mindset Intelligence, Failure and Emotion (PC-SMILE)

SUMMARY:
Depression and anxiety are common mental health problems among adolescents worldwide. In Hong Kong, one in every four secondary school students reports clinical-level depression or anxiety symptoms. Extant research has found that a fixed mindset on intelligence and emotions and failure-is-debilitating belief are closely related to more depression and anxiety symptoms, hopelessness, and suicidality. At the same time, recent research also points to the importance of parental mindset. Parents are the primary social support of adolescents; parental belief systems can strongly influence children's affect, behaviour, and mental health. However, the effects of parent-child mindset interventions on a child's internalising problems have not yet been empirically examined. As emerging evidence has shown the promise of single-session interventions in reducing and preventing youth internalising problems, this project develops and examines a parent and child single-session intervention on mindsets of intelligence, failure, and emotion (PC-SMILE) - to tackle depression and anxiety in young people and promote parental well-being.

Using a three-arm randomised controlled trial, the proposed study will examine the effectiveness of PC-SMILE on reducing depression and anxiety symptoms among children, enhancing well-being and parent-child relationships.

A total of 549 parent-child dyads will be recruited from six secondary schools and randomly assigned to either the PC-SMILE intervention group, the C-SMILE intervention group, or the no-intervention waitlist control group. The intervention is approximately 45 minutes in length. In the PC-SMILE group, both parent and child will receive intervention, and their mental health and family relationship will be assessed at three time points: baseline before intervention (T1), within two weeks post-intervention (T2), and three months post-intervention (T3). In the C-SMILE group, only the child will undergo intervention, while both the child and parent will be required to complete the repeated assessments. A pilot test (n = 9) has supported the feasibility and acceptability of the PC-SMILE intervention. We hypothesise that compared to the waitlist control group, the PC-SMILE intervention group and C-SMILE group will significantly improve child depression and anxiety (primary outcome) and significantly improve secondary outcomes, including children's academic self-efficacy, hopelessness, psychological well-being, and parent-child interactions and relationships, and PC-SMILE group is more effective than C-SMILE group. The intention-to-treat principle and linear-regression-based maximum likelihood multi-level models will be used for data analysis.

As of May 2024, we enrolled 75 students and their parents in the study.

This study will not only provide evidence on parent-child growth mindset intervention for adolescent internalising problems but can also serve as a scalable and accessible intervention for improving the well-being of young people and their parents.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria for adolescent participants are:

  1. aged between 11-16 (inclusive) with one parent willing to participate;
  2. Chinese youth who can read and write in Chinese;
  3. sufficient visual and auditory abilities to complete the intervention and assessment;
  4. ability to give consent to participate in the study.
* The inclusion criteria for parent participants are:

  1. living with the child participant;
  2. Chinese-language proficiency and comfort with completing computer-based activities;
  3. sufficient visual and auditory abilities to complete the intervention and assessment;
  4. ownership of personal internet-equipped devices.

Exclusion Criteria:

* Exclusion criteria for adolescent participants are:

  1. no parental consent;
  2. inability to remain focused to complete the intervention and the survey, which take approximately 45 and 25 minutes respective;
  3. intellectual disability or severe illness or pain that would lead to significant bias in students' health and mental health situation.
* Exclusion criteria for parent participants are:

  1. having a mental illness;
  2. inability to remain focused to complete the intervention and the survey, which take approximately 45 and 25 minutes respective;
  3. intellectual disability or severe illness or pain that would lead to significant bias in students' health and mental health situation.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 549 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Children's depression and anxiety symptoms | baseline
  25-item Revised Children's Anxiety and Depression Scale (RCADS-25)
Children's depression and anxiety symptoms | two weeks post-intervention
  25-item Revised Children's Anxiety and Depression Scale (RCADS-25)
Children's depression and anxiety symptoms | three months post-intervention
  25-item Revised Children's Anxiety and Depression Scale (RCADS-25)

SECONDARY OUTCOMES:
Children's hopelessness | baseline
  the four-item Hopelessness Scale
Children's hopelessness | two weeks post-intervention
  the four-item Hopelessness Scale
Children's hopelessness | three months post-intervention
  the four-item Hopelessness Scale
Children's psychological well-being | baseline
  the Warwick-Edinburgh Mental Well-Being Scale-7
Children's psychological well-being | two weeks post-intervention
  the Warwick-Edinburgh Mental Well-Being Scale-7
Children's psychological well-being | three months post-intervention
  the Warwick-Edinburgh Mental Well-Being Scale-7
Parents' psychological well-being | baseline
  the Warwick-Edinburgh Mental Well-Being Scale-7
Parents' psychological well-being | three months post-intervention
  the Warwick-Edinburgh Mental Well-Being Scale-7
Parent-child relationships | baseline
  three items
Parent-child relationships | two weeks post-intervention
  three items
Parent-child relationships | three months post-intervention
  three items
Parent-child interactions | baseline
  three questions about how many days the children spend more than 15 minutes per day doing activities with their parents in a week
Parent-child interactions | two weeks post-intervention
  three questions about how many days the children spend more than 15 minutes per day doing activities with their parents in a week
Parent-child interactions | three months post-intervention
  three questions about how many days the children spend more than 15 minutes per day doing activities with their parents in a week
Perceived parent learning versus performance orientation | baseline
  8 items for children and 12 items for parents to indicate the extent to which reactions parents would have and which reactions children would perceive
Perceived parent learning versus performance orientation | two weeks post-intervention
  8 items for children and 12 items for parents to indicate the extent to which reactions parents would have and which reactions children would perceive
Perceived parent learning versus performance orientation | three months post-intervention
  8 items for children and 12 items for parents to indicate the extent to which reactions parents would have and which reactions children would perceive
Children's academic self-efficacy | baseline
  a 5-item scale that was adapted from the part of Patterns of Adaptive Learning Survey
Children's academic self-efficacy | two weeks post-intervention
  a 5-item scale that was adapted from the part of Patterns of Adaptive Learning Survey
Children's academic self-efficacy | three months post-intervention
  a 5-item scale that was adapted from the part of Patterns of Adaptive Learning Survey

IPD SHARING:
Plan to Share IPD: No